CLINICAL TRIAL: NCT07020962
Title: The Effect of Laughter Therapy on Distress, Depression and Psychological Well-being in Breast Cancer Patients Before Surgical Intervention: A Randomised Controlled Trial
Brief Title: Effect of Laughter Therapy on Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Servet CİHAN, Education nurse, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ServetCİHAN
Record Dates: First submitted 2025-04-25; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Laughter Therapy; Psychological Well-being; Breast Cancer; Distress; Depression
Keywords: breast cancer; psychological well-being; depression; distress; laughter therapy
MeSH Terms: conditions — Psychological Well-Being; Breast Neoplasms; Depression | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Laughter therapy
  Interventions: Other: laughter therapy
- control group (Active Comparator): routine nursing care
  Interventions: Other: routine nursing care

INTERVENTIONS:
Other: laughter therapy — Laughter therapy/yoga, classified as complementary therapy in medicine, is a unique form of exercise consisting of a combination of laughter, yoga and breathing techniques that allows us to laugh without any sense of humour.
  Arms: Experimental group
Other: routine nursing care — routine nursing care
  Arms: control group

SUMMARY:
The aim of this study is to examine the effect of laughter therapy applied to breast cancer patients before surgical intervention on distress, depression and psychological well-being of patients.

This research will be carried out as an experimental research with a randomised control group.

The population of the study will consist of breast cancer patients diagnosed with breast cancer in a city hospital and scheduled for surgery in the breast-endocrine surgery clinic. The research will be carried out with patients who meet the inclusion criteria and agree to participate in the study. The sample size for the study was calculated using the G* Power 3.1.9.7 programme (Faul et al., 2007). In the calculation, since there was no similar study for two-way mixed design analysis of variance, the required sample size was calculated as 48, 24 in each group, based on the medium effect size (effect size f=0.25), 5% margin of error (alpha=0.05), inter-measurement correlation value 0.5 and 80% power (1-β=0.80). Considering the data losses, the number was increased by 20% and a total of 56 patients in the intervention and control groups constituted the sample of the study.

Hypothesis(es):

H1: The effect of laughter therapy applied to breast cancer patients on distress over time is different in the experimental and control groups.

H2: The effect of laughter therapy applied to breast cancer patients on depression over time is different in the experimental and control groups.

H3: The effect of laughter therapy applied to breast cancer patients on psychological well-being according to time is different in experimental and control groups.

In obtaining the research data; Personal Information Form, Distress Thermometer, Psychological well-being scale prepared by the researchers in line with the literature will be used.

The research data will be collected face-to-face through data collection forms from breast cancer patients diagnosed with breast cancer and scheduled for surgery in the breast-endocrine surgery clinic. Individuals who agree to participate in the study and meet the inclusion criteria will be assigned to the experimental and control groups by providing randomisation. Which caregivers will be in the intervention group and which will be in the control group will be determined according to the randomisation table determined by https://www.randomizer.org/ over the internet. Group 1: Intervention Group, Group 2: Control Group. Data collection tools will be applied to the individuals in the experimental and control groups as a pre-test. Individuals in the experimental group will receive laughter therapy three days a week for 30-45 minutes (6 sessions). Individuals in the control group will receive only standard nursing care. Data collection tools will be applied to the individuals in both groups for post-test, 1 and 3-month follow-up tests immediately after all laughter sessions with the experimental group are completed.

DETAILED DESCRIPTION:
Breast cancer is described as a type of disease caused by the uncontrolled proliferation of cells surrounding the milk glands and ducts in the breast. Breast cancer is the most common type of cancer in women in the world and in our country. According to GLOBOCAN 2022 data, breast cancer constitutes 23.8% of all female cancers, and it was reported that 2.3 million women worldwide and 25 thousand women in Turkey were diagnosed with breast cancer in 2022.

As a result of mastectomy or breast conserving treatment, breast cancer can bring about various negative consequences such as body image and sexual life disorder. Women diagnosed with breast cancer often experience psychological problems such as fear of cancer recurrence, deterioration of body perception, decreased self-esteem, loss of femininity and fear of death, and cancer diagnosis and treatment can lead to anxiety, depression and anger in patients. Studies have reported that diagnosis, treatment outcomes, and the course of the disease are associated with depressive symptoms .Depressive symptoms have been identified as one of the most common complications in patients with breast cancer. Depression and anxiety are common diagnoses following breast cancer diagnosis and are vital as effective ways to identify patients at risk for psychological distress.

Psychosocial distress has long been identified as an important problem for breast cancer patients who face challenges in many different areas. The National Comprehensive Cancer Network (NCCN) has recognised distress as an important sequela of cancer diagnosis and treatment. In a qualitative study examining the preoperative distress and anxiety experiences of breast cancer patients, it was reported that the anxiety and distress of these patients increased mostly before surgery, but they were also affected by the care experiences surrounding their surgery. Formally, cancer-related distress is defined as 'a multifactorial unpleasant emotional experience of a psychological (i.e. cognitive, behavioural, emotional), social or spiritual nature that may interfere with the ability to cope effectively with cancer, its physical symptoms and treatment'. In addition, the definition of distress has drawn attention to the early identification and treatment of emotional distress in cancer, and the conceptualisation of psychological distress as the 6th vital sign has provided a framework for care providers to understand emotional difficulties in cancer patients. In a systematic review, it was reported that unmanaged distress negatively affects cancer-related morbidity and mortality as well as quality of life.

The diagnosis and treatment process of breast cancer may increase the level of depression and psychological distress and have a negative impact on the psychological well-being of patients. Psychological well-being is defined as the individual's self-actualisation, using his/her existing or unrealised potential in the most efficient way, accepting himself/herself with this potential, having life goals, establishing qualified relationships and feeling responsibility for his/her own life . It is stated that individuals with high levels of psychological well-being not only feel good about themselves, but also are more successful in interpersonal relationships, their life energy and creativity increase, their immune systems are strengthened, and they are more productive in business life. In the light of this information, considering that having cancer is one of the most stressful life events, psychological well-being levels should be increased in order to overcome the negative consequences of being diagnosed with breast cancer.

In recent years, laughter therapy has attracted attention among methods of coping with stress. Laughter therapy/yoga, which is classified as complementary therapy in medicine, is a unique form of exercise consisting of a combination of laughter, yoga and breathing techniques that allow us to laugh without any sense of humour. Although it is a different approach from other therapeutic methods, it focuses on the approach that both body and mind can only be healthy when the psychological aspects of the brain change. Laughter yoga can be used as a nursing intervention to reduce the symptoms of different diseases and relieve general stress. Laughter yoga has been registered by the NIC (classification of nursing interventions) authority at the University of Iowa since 2023 and has been included in the latest version of the NIC. In this context, it is envisaged that laughter yoga as a nursing initiative will be widely used in nursing research and education in caring for both sick and healthy individuals.

It is reported that humour and laughter yoga are humane, allow the improvement of the experience in the hospital environment, and contribute to the development of communication and trust between the nurse and the individual while providing care. In addition, it enables the person to participate in care and treatment, helps to increase comfort, helps to cope with difficult and unpleasant situations, reduces anger, tension, stress, increases the person's tolerance to pain, and strengthens the immune system.

As a result of a systematic review and metanalysis, it was suggested that nurses should actively transform this therapy into clinical practice to alleviate the negative emotions of patients and teach these methods to patients and their relatives as part of health education to improve treatment outcomes. In the same study, it was concluded that laughter yoga is a multimodality flexible therapy suitable for improving the negative emotions of cancer patients. However, it is stated that in order to evaluate the effect of laughter therapy on patient outcomes in cancer patients, studies with larger samples, different cancer types, long-term follow-ups, and more randomised controlled designs should be conducted. It was also stated that more studies are needed to show whether laughter therapy reduces depressive symptoms in cancer patients.

It is also recommended that future studies try to obtain more precise results regarding the effect of laughter therapy by extending the intervention time in cancer patients.

It is a very exciting and innovative practice for nurses to use laughter yoga to protect and improve the health of individuals. In our country, a limited number of studies have been conducted on laughter yoga, which has become increasingly widespread and its benefits have been scientifically approved. In addition, no study has been found in our country that examines the effect of laughter therapy on the distress, depression and psychological well-being levels of patients before the surgical procedure in breast cancer patients. Considering the gaps in the literature, this study aimed to investigate the effect of laughter therapy applied to breast cancer patients before surgical intervention on distress, depression and psychological well-being levels of patients in a randomised controlled longitudinal study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary acceptance to participate in the study,
* Being diagnosed with breast cancer and being in the patient group in which surgical operation is planned,
* Not having participated in laughter yoga practice before,
* Being literate,
* Not having a psychiatric disease (diagnosis)
* Not having a communication and understanding disability related to vision, hearing
* Being in the age group of 18 and over

Exclusion Criteria:

* Not wanting to participate in the study,
* Being in the patient group with a condition recommended not to do laughter yoga (having undergone surgery in the abdominal region in the last three months, uncontrolled hypertension, glaucoma, hernia, epilepsy),
* Not having participated in any of the laughter yoga sessions,
* Having physical restriction/respiratory problems and not being able to perform yoga movements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Laughter therapy will be applied to individuals with breast cancer and their levels of psychological distress will be measured.Laughter therapy will be applied to individuals with breast cancer and their psychological distress levels will be measured. | 2 weeks
  Meme kanserine sahip olan bireylere kahkaha terapisi uygulanacak ve pskilojik sıkıntı düzeyleri ölçülecektir.
  Laughter therapy will be applied to individuals with breast cancer and their levels of psychological distress will be measured. (Face to face training will be given)
Laughter therapy will be applied to individuals with breast cancer and their depression levels will be measured. | 2 weeks
  Laughter therapy will be applied to individuals with breast cancer and their depression levels will be measured (Face to face training will be given)
Laughter therapy will be applied to individuals with breast cancer and their psychological well-being levels will be measured. | 2 weeks
  Laughter therapy will be applied to individuals with breast cancer and their psychological well-being levels will be measured (Face to face training will be given)

CONTACTS AND LOCATIONS:
Overall Officials: Servet Cihan, Principal Investigator — Prof. Dr. Cemil Taşcıoğlu Şehir Hastanesi

IPD SHARING:
Plan to Share IPD: No